CLINICAL TRIAL: NCT03340688
Title: Cervical Cerclage for Preventing Spontaneous Preterm Birth in Twin Pregnancies With Transvaginal Ultrasound Cervical Length ≤ 15mm: a Study Protocol for a Randomized Clinical Trial
Brief Title: Cerclage for Twins With Short Cervical Length ≤ 15mm
Acronym: TWIN-UIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Collaborators: Federico II University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17D.326
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Twin Pregnancy With Antenatal Problem; Preterm Birth; Short Cervix
MeSH Terms: conditions — Premature Birth | interventions — Cerclage, Cervical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical cerclage + vaginal progesterone (Active Comparator): Cervical cerclage in twin pregnancy with transvaginal cervical length ≤15mm and Daily vaginal progesterone 400mg from diagnosis of short cervix to 36 weeks
  Interventions: Procedure: Cervical cerclage
- Vaginal progesterone (No Intervention): Daily vaginal progesterone 400mg from diagnosis of short cervix to 36 weeks

INTERVENTIONS:
Procedure: Cervical cerclage — Cervical cerclage indicated by short cervix ≤15mm
  Arms: Cervical cerclage + vaginal progesterone

SUMMARY:
This is a multicenter randomized study designed to determine if ultrasound indicated cerclage reduces the incidence of spontaneous preterm birth <34 weeks in asymptomatic women with twin gestations and cervical length ≤15mm, diagnosed by transvaginal ultrasound between 16 to 23 6/7 weeks of gestation.

DETAILED DESCRIPTION:
Twin pregnancies have 59% incidence of preterm delivery (before 37 weeks of gestation), with increased perinatal mortality and neonatal morbidity. No therapy has proven effective in preventing preterm birth in twins. The transvaginal cervical length (TVCL) performed before 24 weeks have been determined to be the best tool to identified women with twin pregnancy at risk of preterm birth (PTB). When short TVCL is identified before 24 weeks, the risk of preterm birth is 60%-70% for TVCL ≤25mm and 80%-90% for TVCL ≤15mm. There are a small number of case reports of cervical cerclage in twin pregnancies with cervical length ≤15mm that suggest decreased preterm birth by 80%. The investigators' objective is to determine if ultrasound indicated cerclage in reduces the incidence of spontaneous preterm birth <34 weeks and improve perinatal outcome in asymptomatic women with twin gestations and cervical length ≤15mm between 16 to 23 6/7 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women more than 18 years of age (limits the participants to female gender)
2. Diamniotic twin pregnancy
3. Asymptomatic
4. Transvaginal cervical length ≤ 15 mm between 16-23 6/7 weeks gestation

Exclusion Criteria:

1. Singleton or higher order than twins multiple gestation
2. Transvaginal cervical length >15mm
3. Cervical dilation with visible amniotic membranes
4. Amniotic membranes prolapsed into the vagina
5. Fetal reduction after 14 weeks form higher order
6. Monoamniotic twins
7. Twin-twin transfusion syndrome
8. Ruptured membranes
9. Major fetal structural anomaly
10. Fetal chromosomal abnormality
11. Cerclage already in place for other indication
12. Active vaginal bleeding
13. Clinical chorioamnionitis
14. Placenta previa
15. Painful regular uterine contractions
16. Labor

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only pregnant women
Enrollment: 200 (Estimated)
Dates: Start 2017-06-22 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Preterm delivery less than 34 weeks | at delivery
  Incidence of preterm birth less than 34 weeks (any indication)

SECONDARY OUTCOMES:
Spontaneous preterm birth rates | at delivery
  Incidence of spontaneous preterm birth less than 34 weeks
Preterm delivery less than <32 weeks, <28 weeks, or <24 weeks | at delivery
  Incidence of preterm birth less than <32 weeks, <28 weeks, or <24 weeks
Mean gestational age at delivery | at delivery
  Mean value of gestational age at delivery (weeks)
Birth weight at birth | at delivery
  Mean value (grams)
Gestational age at spontaneous rupture of membranes | at delivery
  Mean value (weeks) through study completion
Premature rupture of membranes | at delivery
  Incidence
Chorioamnionitis | at delivery
  Incidence
Composite adverse neonatal outcome | Incidence between birth and 28 days of age
  Includes necrotizing enterocolitis, intraventricular hemorrhage (grade 3 or higher), respiratory distress syndrome, bronchopulmonary dysplasia, retinopathy, blood-culture proven sepsis
Neonatal death | Between birth and 28 days of age
  Incidence
Maternal death | Between birth and 6 weeks postpartum
  Incidence
Interval between diagnosis and delivery | at delivery
  Mean value (days) through study completion

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Roman, MD, Principal Investigator — Thomas Jefferson University
Locations (8):
- United States (3):
  - George Washington University, Washington D.C., District of Columbia
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Austin Maternal Fetal Medicine St David's Health Care, Austin, Texas
- The Egyptian IVF Center, Cairo, Egypt
- Italy (3):
  - Bologna University, Bologna
  - University of Brescia, Brescia
  - Università degli Studi di Napoli "Federico II", Naples
- University of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Result] Hamilton BE, Hoyert DL, Martin JA, Strobino DM, Guyer B. Annual summary of vital statistics: 2010-2011. Pediatrics. 2013 Mar;131(3):548-58. doi: 10.1542/peds.2012-3769. Epub 2013 Feb 11. PMID 23400611
- [Result] Goldenberg RL, Iams JD, Miodovnik M, Van Dorsten JP, Thurnau G, Bottoms S, Mercer BM, Meis PJ, Moawad AH, Das A, Caritis SN, McNellis D. The preterm prediction study: risk factors in twin gestations. National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Am J Obstet Gynecol. 1996 Oct;175(4 Pt 1):1047-53. doi: 10.1016/s0002-9378(96)80051-2. PMID 8885774
- [Result] Conde-Agudelo A, Romero R, Hassan SS, Yeo L. Transvaginal sonographic cervical length for the prediction of spontaneous preterm birth in twin pregnancies: a systematic review and metaanalysis. Am J Obstet Gynecol. 2010 Aug;203(2):128.e1-12. doi: 10.1016/j.ajog.2010.02.064. Epub 2010 Jun 23. PMID 20576253
- [Result] Saccone G, Rust O, Althuisius S, Roman A, Berghella V. Cerclage for short cervix in twin pregnancies: systematic review and meta-analysis of randomized trials using individual patient-level data. Acta Obstet Gynecol Scand. 2015 Apr;94(4):352-8. doi: 10.1111/aogs.12600. Epub 2015 Mar 1. PMID 25644964
- [Result] Roman A, Rochelson B, Fox NS, Hoffman M, Berghella V, Patel V, Calluzzo I, Saccone G, Fleischer A. Efficacy of ultrasound-indicated cerclage in twin pregnancies. Am J Obstet Gynecol. 2015 Jun;212(6):788.e1-6. doi: 10.1016/j.ajog.2015.01.031. Epub 2015 Jan 28. PMID 25637840
- [Result] Romero R, Conde-Agudelo A, El-Refaie W, Rode L, Brizot ML, Cetingoz E, Serra V, Da Fonseca E, Abdelhafez MS, Tabor A, Perales A, Hassan SS, Nicolaides KH. Vaginal progesterone decreases preterm birth and neonatal morbidity and mortality in women with a twin gestation and a short cervix: an updated meta-analysis of individual patient data. Ultrasound Obstet Gynecol. 2017 Mar;49(3):303-314. doi: 10.1002/uog.17397. PMID 28067007

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT03340688/Prot_SAP_000.pdf
  • Informed Consent Form (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT03340688/ICF_001.pdf